CLINICAL TRIAL: NCT01504412
Title: An Asian, Phase 2, Multicenter, Randomized, Double-blind, Placebo- and Pregabalin-controlled, Dose-finding Study of DS-5565 in Patients With Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Asian Phase 2 Study for Treatment of Pain Associated With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS5565-A-J202
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Pain; Diabetic Peripheral Neuropathy
Keywords: Pain; Diabetic Peripheral Neuropathy
MeSH Terms: conditions — Pain | interventions — mirogabalin; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- DS-5565 Low Dose (Experimental): DS-5565 10mg/day, administered in 2 doses. Treatment period: 1 week titration and 6 weeks of fixed dose.
  Interventions: Drug: DS-5565
- DS-5565 Middle Dose (Experimental): DS-5565 20mg/day, administered in 2 doses. Treatment period: 1 week titration and 6 weeks of fixed dose.
  Interventions: Drug: DS-5565
- DS-5565 High Dose (Experimental): DS-5565 30mg/day, administered in 2 doses. Treatment period: 1 week titration and 6 weeks of fixed dose.
  Interventions: Drug: DS-5565
- Placebo (Placebo Comparator): DS-5565 placebo oral tablets and pregabalin placebo oral capsules administered 2 times per day.
  Interventions: Drug: Placebo
- Pregabalin (Active Comparator): Pregabalin capsules 300mg/day administered in 2 doses
  Interventions: Drug: Pregabalin capsules

INTERVENTIONS:
Drug: DS-5565 — Oral tablets administered twice daily
  Arms: DS-5565 Low Dose
Drug: DS-5565 — Oral tablets administered twice daily
  Arms: DS-5565 Middle Dose
Drug: DS-5565 — Oral tablets administered twice daily
  Arms: DS-5565 High Dose
Drug: Placebo — DS-5565 placebo oral tablets and pregabalin placebo oral capsules administered 2 times per day
  Arms: Placebo
Drug: Pregabalin capsules — Pregabalin oral capsules 150 mg administered twice a day
  Arms: Pregabalin

SUMMARY:
The purpose of this study is to investigate the effectiveness and safety of DS-5565, compared to placebo, in subjects with pain associated with diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes mellitus
* Painful distal symmetric polyneuropathy
* Average daily pain score is great than or equal to 4

Exclusion Criteria:

* HbA1c greater than 9.0

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Tokyo, Japan
- Seoul, South Korea
- Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Baba M, Kuroha M, Ohwada S, Murayama E, Matsui N. Results of Mirogabalin Treatment for Diabetic Peripheral Neuropathic Pain in Asian Subjects: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Study. Pain Ther. 2020 Jun;9(1):261-278. doi: 10.1007/s40122-020-00156-6. Epub 2020 Feb 12. PMID 32052264

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met all inclusion criteria and none of the exclusion criteria were enrolled and randomized to treatment.
Pre-assignment Details: Enrolled participants were equally randomized (1:1:1:1:1) to placebo, pregabalin, or one of three different doses of DS-5565 in a double-blind fashion. After randomization, participants received one-half the fixed dose for the first week, and subsequently received the fixed dose for 6 weeks. All participants were followed for an additional week.
Groups:
- Pregabalin: Pregabalin capsules 300 mg/day administered in 2 doses
- DS-5565 10 mg/Day: DS-5565 10 mg/day, administered in 2 doses (5 mg twice daily).
- DS-5565 20 mg/Day: DS-5565 20 mg/day, administered in 2 doses (10 mg twice daily).
- DS-5565 30 mg/Day: DS-5565 30mg/day, administered in 2 doses (15 mg twice daily).
Period: Overall Study
Arm/Group | Placebo | Pregabalin | DS-5565 10 mg/Day | DS-5565 20 mg/Day | DS-5565 30 mg/Day
Started | 89 | 87 | 90 | 94 | 90
Completed | 84 | 75 | 86 | 75 | 77
Not Completed | 5 | 12 | 4 | 19 | 13
Not completed — Adverse Event | 1 | 8 | 1 | 7 | 10
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 5 | 1
Not completed — Other | 2 | 1 | 1 | 6 | 1
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin | DS-5565 10 mg/Day | DS-5565 20 mg/Day | DS-5565 30 mg/Day | Total
Number analyzed (Participants) | 89 | 87 | 90 | 94 | 90 | 450
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 64 | 61 | 56 | 60 | 69 | 310
  >=65 years | 25 | 26 | 34 | 34 | 21 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.79) | 60.1 (8.74) | 60.5 (9.77) | 60.9 (9.32) | 59.0 (10.06) | 59.8 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 31 | 36 | 41 | 160
  Male | 62 | 62 | 59 | 58 | 49 | 290
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 89 | 87 | 90 | 94 | 90 | 450
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 89 | 87 | 90 | 94 | 90 | 450
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Average Daily Pain Score From Baseline Among Participants Who Received DS5565 for Pain Associated With Diabetic Peripheral Neuropathy
Description: The mean change in average daily pain score (ADPS) was measured using a 11-point numeric rating scale (NRS; 0 [no pain] to 10 [worst possible pain]. The rating averaged over a 7-day period and was based on entries in patients' daily pain diaries. Greater mean changes (improvements) in ADPS indicated better outcomes. A minimally meaningful effect was a mean decrease of at least 1.0 point [scale of 0 to 10] versus placebo.
Time Frame: Baseline to Week 7 postdose
Population: Mean change in ADPS was assessed in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin | DS-5565 10 mg/Day | DS-5565 20 mg/Day | DS-5565 30 mg/Day
Number analyzed (Participants) | 88 | 85 | 90 | 93 | 90
units on a scale
  Baseline to Week 1 | -0.59 (1.13) | -0.71 (1.29) | -0.69 (0.90) | -0.88 (1.32) | -0.60 (1.01)
  Baseline to Week 2 | -0.86 (1.36) | -0.92 (1.33) | -1.16 (1.06) | -1.21 (1.56) | -1.06 (1.28)
  Baseline to Week 3 | -1.05 (1.38) | -1.06 (1.29) | -1.32 (1.15) | -1.50 (1.68) | -1.35 (1.52)
  Baseline to Week 4 | -1.12 (1.47) | -1.29 (1.48) | -1.50 (1.22) | -1.65 (1.68) | -1.56 (1.53)
  Baseline to Week 5 | -1.28 (1.62) | -1.44 (1.56) | -1.62 (1.32) | -1.68 (1.80) | -1.47 (1.61)
  Baseline to Week 6 | -1.41 (1.68) | -1.40 (1.51) | -1.79 (1.31) | -1.78 (1.68) | -1.68 (1.50)
  Baseline to Week 7 | -1.50 (1.77) | -1.55 (1.77) | -1.82 (1.36) | -1.91 (1.77) | -1.75 (1.68)
Statistical Analysis 1: Comparison: Placebo vs DS-5565 10 mg/Day; Test type: Superiority; p = 0.1995, ANCOVA — Dunnett method was used for adjustment of multiple testing; Hazard Ratio (HR) = -0.42, 95% CI 2-sided [-0.99 to 0.15]
Statistical Analysis 2: Comparison: Placebo vs DS-5565 20 mg/Day; Test type: Superiority; p = 0.2886, ANCOVA — Dunnett method was used for adjustment of multiple testing; Hazard Ratio (HR) = -0.37, 95% CI 2-sided [-0.93 to 0.20]
Statistical Analysis 3: Comparison: Placebo vs DS-5565 30 mg/Day; Test type: Superiority; p = 0.4704, ANCOVA — Dunnett method was used for adjustment of multiple testing; Hazard Ratio (HR) = -0.30, 95% CI 2-sided [-0.87 to 0.27]

2. Secondary Outcome: Mean Change in Short Form-McGill Pain Questionnaire From Baseline Among Participants Who Received DS5565 for Pain Associated With Diabetic Peripheral Neuropathy
Description: The Short Form-McGill Pain Questionnaire (SF-MPQ) Visual Analog Scale (VAS) is reported. For VAS, participants rated pain intensity on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain.
  Greater mean changes (improvements) in SF-MPQ indicated better outcomes.
Time Frame: at Week 7 postdose
Population: Mean change in SF-MPQ VAS was assessed in the Full Analysis Set.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin | DS-5565 10 mg/Day | DS-5565 20 mg/Day | DS-5565 30 mg/Day
Number analyzed (Participants) | 88 | 85 | 90 | 93 | 90
units on a scale | -16.7 (2.03) | -17.2 (2.06) | -21.9 (2.01) | -22.1 (1.97) | -24.2 (2.00)
Statistical Analysis 1: Comparison: Placebo vs DS-5565 10 mg/Day; This analysis assessed placebo vs DS-5565 10 mg/day for the visual analog scale; Test type: Superiority; p = 0.0691, ANCOVA; Least squares mean difference = -5.2, 95% CI 2-sided [-10.8 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs DS-5565 20 mg/Day; This analysis assessed placebo vs DS-5565 20 mg/day for the visual analog scale; Test type: Superiority; p = 0.0577, ANCOVA; Least squares mean difference = -5.4, 95% CI 2-sided [-10.9 to 0.2]
Statistical Analysis 3: Comparison: Placebo vs DS-5565 30 mg/Day; This analysis assessed placebo vs DS-5565 30 mg/day for the visual analog scale; Test type: Superiority; p = 0.0093, ANCOVA; Least squares mean difference = -7.4, 95% CI 2-sided [-13.0 to -1.8]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time the Informed Consent Form was signed to 7 days after the last dose of study medication, approximately 18 months.
Description: Adverse events that appeared for the first time during treatment, or that worsened relative to the pre-treatment state, were analyzed. Additionally, 3 participants who had major violations of GCP were excluded from the Safety Analysis Set (1 participant each in the placebo, pregabalin, and in the 20-mg/day group).
Groups:
- DS-5565 10 mg/Day: DS-5565 10 mg/day, administered in 2 doses (5 mg twice daily). Treatment period: 1 week titration and 6 weeks of fixed dose.
- DS-5565 20 mg/Day: DS-5565 20 mg/day, administered in 2 doses (10 mg twice daily). Treatment period: 1 week titration and 6 weeks of fixed dose.
- DS-5565 30 mg/Day: DS-5565 30mg/day, administered in 2 doses (15 mg twice daily). Treatment period: 1 week titration and 6 weeks of fixed dose.
Arm/Group | Placebo | Pregabalin | DS-5565 10 mg/Day | DS-5565 20 mg/Day | DS-5565 30 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/86 | 0/90 | 1/93 | 0/90
Serious Adverse Events (participants affected / at risk) | 3/88 | 2/86 | 1/90 | 4/93 | 2/90
Other Adverse Events (participants affected / at risk) | 13/88 | 28/86 | 18/90 | 38/93 | 42/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=88) | Pregabalin (N=86) | DS-5565 10 mg/Day (N=90) | DS-5565 20 mg/Day (N=93) | DS-5565 30 mg/Day (N=90)
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Metastases to lymph node (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=88) | Pregabalin (N=86) | DS-5565 10 mg/Day (N=90) | DS-5565 20 mg/Day (N=93) | DS-5565 30 mg/Day (N=90)
Nasopharyngitis (Infections and infestations) | 3 | 2 | 7 | 13 | 3
Somnolence (Nervous system disorders) | 5 | 12 | 8 | 13 | 19
Dizziness (Nervous system disorders) | 3 | 9 | 5 | 10 | 15
Headache (Nervous system disorders) | 2 | 5 | 2 | 4 | 3
Vomiting (Gastrointestinal disorders) | 1 | 5 | 1 | 3 | 2
Oedema peripheral (General disorders) | 1 | 5 | 3 | 3 | 7
Gait disturbance (General disorders) | 1 | 4 | 1 | 7 | 2
Weight increased (Investigations) | 0 | 2 | 1 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No